CLINICAL TRIAL: NCT02950922
Title: Study of RVT-501 in Adult and Adolescent Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dermavant Sciences GmbH (Industry)
Responsible Party: Sponsor
Organization: Dermavant Sciences, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVT-501-2001
Record Dates: First submitted 2016-10-11; First posted 2016-11-01 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — methyl 4-(((3-(6,7-dimethoxy-2-(methylamino)quinazolin-4-yl)phenyl)amino)carbonyl)benzoate; Ointments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- RVT-501 0.2% ointment (Experimental): RVT-501 0.2% ointment BID x 28 days (30 adults, 20 adolescents)
  Interventions: Drug: RVT-501 0.2% ointment
- RVT-501 0.5% ointment (Experimental): RVT-501 0.5% ointment BID x 28 days (30 adults, 20 adolescents)
  Interventions: Drug: RVT-501 0.5% ointment
- Vehicle ointment (Placebo Comparator): Vehicle ointment BID x 28 days (30 adults, 20 adolescents)
  Interventions: Other: Vehicle ointment

INTERVENTIONS:
Drug: RVT-501 0.2% ointment
  Arms: RVT-501 0.2% ointment
Drug: RVT-501 0.5% ointment
  Arms: RVT-501 0.5% ointment
Other: Vehicle ointment — Placebo comparator
  Arms: Vehicle ointment

SUMMARY:
This is a multi-center, randomized, vehicle-controlled, double-blind Phase 2 study in adults and adolescent subjects with mild to moderate atopic dermatitis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, efficacy, and pharmacokinetics of the 0.2% BID and 0.5% concentrations of RVT-501 in patients with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Males and females with confirmed diagnosis of atopic dermatitis by Hanifin and Rajka criteria (Appendix 4: Criteria for Atopic Dermatitis Diagnosis).

   For adult subjects, the age range is 18 to 70 years. For adolescent subjects, the age range is 12 to 17 years.
2. Subjects with atopic dermatitis covering ≥ 3% and < 40% of the body surface area and with an Investigator Global Assessment (IGA) of 2 or 3 (mild to moderate) at baseline. Scalp, palms and soles should be excluded from the BSA calculation to determine eligibility at baseline.

   NOTE: Subjects with mild disease (IGA =2) will be limited to approximately 25% of total enrollment.
3. Minimum EASI score of 7 at baseline.
4. Females of childbearing potential and male subjects and who are engaging in sexual activity that could lead to pregnancy must use the following adequate birth control methods while on study and for 2 weeks after stopping study drug. Acceptable contraception methods are:

   * Male or Male partner with vasectomy OR
   * Male condom, AND partner use of one of the contraceptive options below:
   * Spermicide
   * Contraceptive subdermal implant that meets effectiveness criteria including a <1% rate of failure per year, as stated in the product label
   * Intrauterine device or intrauterine system that meets effectiveness criteria including a <1% rate of failure per year, as stated in the product label [Hatcher, 2007a]
   * Oral Contraceptive, either combined or progestogen alone [Hatcher, 2007a] Injectable progestogen [Hatcher, 2007a]
   * Contraceptive vaginal ring [Hatcher, 2007a]
   * Percutaneous contraceptive patches [Hatcher, 2007a]

   These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

   Non-child-bearing potential is defined as pre-menopausal females with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy; hysteroscopic sterilization; or postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40mlU is confirmatory. Documented verbal history from the subject is acceptable.
5. Atopic Dermatitis present for at least 12 months according to the patient/care giver and stable disease for at least 1 month according to the patient/care giver.
6. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

-

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. A positive Hepatitis B surface antigen or positive Hepatitis C antibody result at screening.
2. A positive test for human immunodeficiency virus (HIV) antibody at screening.
3. Screening alanine aminotransferase (ALT) ≥ 3x the upper limit of normal (ULN).
4. Total bilirubin > 1.5x the upper limit of normal (ULN); total bilirubin > ULN and ≤ 1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%.
5. Corrected QT (QTc) interval >475 msec or >525 msec in the presence of bundle branch block.
6. Subjects with a present illness of Kaposi's varicelliform eruption, scabies, molluscum contagiosum, impetigo, psoriasis, connective tissue disorder, or Netherton's syndrome, or any other disease which could have an effect on the pathological evaluation of atopic dermatitis.
7. Use of any prohibited medication.

   Prohibited concomitant medications, therapy, etc. during the defined period are as follows. If a subject requires any of these medications throughout the study period, he/she may be excluded from or discontinued from the study, at the discretion of the investigator and medical monitor.

   From 6 months prior to the first application of study drugs to the completion of the follow-up examination or discontinuation:
   * Biological products that might have significantly affected the evaluation of atopic dermatitis condition (e.g., TNF inhibitors, anti-IgE antibodies, anti-CD20 antibodies, anti-IL4 receptor)

   From 28 days prior to the first application of study drug until the completion of the Treatment Phase or discontinuation:
   * Corticosteroid preparations (oral, injection, and suppository preparations) and topical corticosteroids that were classified as super high potency (clobetasol propionate). Eye drop and nasal preparations are allowed. Inhaled preparations are allowed if used for a stable condition and at a stable dose for > 28 days before screening, and are continued at the same dose throughout the study.
   * Oral preparations and injections of immunosuppressants (cyclosporine, methotrexate, azathioprine, tacrolimus, etc.)
   * Over the counter or herbal medicines for atopic dermatitis (topical and oral preparations)
   * Excessive sun exposure, tanning booth, other UV light source and phototherapy including PUVA therapy

   From 7 days prior to the first application of the study drugs to the completion of the Treatment Phase or discontinuation:
   * Topical corticosteroids that were classified as low, medium, or high potency (fluocinonide, triamcinolone acetonide, desonide, hydrocortisone). Eye drop and nasal preparation are allowed.
   * Tacrolimus and pimecrolimus cream and/or ointment
   * Antihistamines/anti-allergics (oral, topical and injections): diphenhydramine, chlorpheniramine maleate, hydroxyzine).

   NOTE: The following antihistamines are allowed:
   * Loratadine, fexofenadine hydrochloride, cetirizine hydrochloride

   From baseline throughout the treatment period
8. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
9. Pregnant females as determined by positive serum (screening) or urine (baseline) human chorionic gonadotropin test at screening or prior to dosing.
10. Lactating females.
11. History of sensitivity to the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
12. The subject has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
13. Current or a history of cancer within 5 years with the exception of fully excised skin basal cell carcinoma, squamous cell carcinoma or carcinoma in situ of the cervix.
14. Subjects with active infection that required oral or intravenous administration of antibiotics, antifungal or antiviral agents within 7 days of Baseline/Day 0.
15. Concurrent skin lesions in the treatment area or pruritus due to conditions other than atopic dermatitis that, in the opinion of the investigator, would either interfere with study evaluations or affect the safety of the subject.
16. Subjects with advanced disease or abnormal laboratory test values that could affect the safety of the subject or the implementation of this study.
17. Evidence of significant hepatic, renal, respiratory, endocrine, hematologic, neurologic, psychiatric, or cardiovascular system abnormalities or laboratory abnormality that will affect the health of the subject or interfere with interpretation of the results.
18. The subject has excessive sun exposure, is planning a trip to a sunny climate which would involve excessive sun exposure, or used tanning booths within 28 days prior to baseline (Day 0) or is not willing to minimize natural and artificial sunlight exposure during the study.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2016-11; Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of adverse events (local and systemic) | 28 days
  Adverse events will be coded using the most current release of MedDRA® (Medical Dictionary for Regulatory Activities). The number and proportion of subjects with adverse events will be summarized by treatment, system organ class, and preferred term for all adverse events, all adverse events considered by the investigator to be related to study drug, all serious adverse events, and all adverse events leading to study drug discontinuation
Laboratory values | 28 days
  Selected laboratory data will be summarized by the observed data and by the change from baseline (as appropriate) across time. Incidence of treatment emergent laboratory values that are considered clinically significantly abnormal will be summarized by treatment group.
Vital signs | 28 days
  Vital signs will be measured in supine or semi-supine position after a 5 minute rest and will include systolic and diastolic blood pressure and pulse rate. Vital sign data will be listed by subject and summarized by treatment.
ECGs | 28 Days
  Single 12-lead ECGs will be obtained at Screening, Day 0, Day 7, Day 28 and during follow up 7-10 days-post-dose using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals. ECG data will be listed by subject and summarized by treatment.
Plasma concentrations of RVT-501 | 28 Days
  PK samples will be collected pre-dose at week 1 for all subjects. At week 4, PK samples will be collected pre-dose and within 2-4 hours post-dose. RVT-501 will be measured in plasma by validated assay in all subjects to confirm exposure. These plasma concentrations will be listed separately for adults and adolescents by metabolite, subject, treatment, and time; and will be summarized by metabolite, treatment and time. The number of percent of subjects with measurable concentration at each time point and any time during the study will be provided.
Plasma concentrations of M11 metabolite | 28 Days
  PK samples will be collected pre-dose at week 1 for all subjects. At week 4, PK samples will be collected pre-dose and within 2-4 hours post-dose. The M11 metabolite will be measured in plasma by validated assay in all subjects to confirm exposure. These plasma concentrations will be listed separately for adults and adolescents by metabolite, subject, treatment, and time; and will be summarized by metabolite, treatment and time. The number of percent of subjects with measurable concentration at each time point and any time during the study will be provided.

SECONDARY OUTCOMES:
Efficacy - Investigators Global Assessment (IGA) | 28 days
  The Investigator's Global Assessment (IGA) of Disease Severity will be assessed at every on-site study visit. The IGA is a global assessment of the current state of the disease. It is a 5-point morphological assessment of overall disease severity All efficacy analyses will be performed based on the ITT population by treatment and age group. The total IGA scores, changes and percent changes from baseline will be summarized by treatment group and visit. The between treatment comparisons will be performed using an ANCOVA model similar to the model used for the EASI score
Efficacy - Eczema Area and Severity Index (EASI) | 28 Days
  The Eczema Area and Severity Index (EASI) will be assessed at every study visit. It quantifies the severity of a subject's atopic dermatitis based on both lesion severity and the percent of BSA affected. The total and regional EASI scores will be summarized for the actual, change from baseline and percent change from baseline. The between treatment comparisons of change and percent change from baseline will be performed by visit using an analysis of covariance model (ANCOVA)
Efficacy - Numeric Rating Scale (NRS) for Pruritus | 28 Days
  NRS for Pruritus (Numerical Rating Scale) is a validated scale used to quickly assess pruritus severity. The total affected BSA and NRS for Pruritus will be analyzed similar to the EASI score. The patient reported symptoms and outcomes will be listed and summarized

OTHER OUTCOMES:
Patient Reported Symptoms | 28 days
  The subject will assess burning and pruritus at the application site during clinic visits on a scale of (0) None to (3) Severe. The patient reported symptoms and outcomes will be listed and summarized.
Patient Report Outcomes | 28 Days
  The Patient Oriented Eczema Measures (POEM - adult version) is a tool used for monitoring atopic dermatitis severity. It focuses on the illness as experienced by the patients. Measurements will be assessed on Day 0, Day 28 and during follow up 7-10 days post dose. The patient reported symptoms and outcomes will be listed and summarized

CONTACTS AND LOCATIONS:
Overall Officials: James Lee, MD, PhD, Study Chair — Dermavant Sciences, Chief Medical Officer
Locations (17):
- United States (13):
  - Dermavant Investigator Site, Fremont, California
  - Dermavant Investigator Site, Los Angeles, California
  - Dermavant Investigator Site, San Diego, California
  - Dermavant Investigator Site, San Luis Obispo, California
  - Dermavant Investigator Site, Louisville, Kentucky
  - Dermavant Investigator Site, Berlin, New Jersey
  - Dermavant Investigator Site, Portland, Oregon
  - Dermavant Investigator Site, Hershey, Pennsylvania
  - Dermavant Investigator Site, Johnston, Rhode Island
  - Dermavant Investigational Site, Dallas, Texas
  - Dermavant Investigator Site, Houston, Texas
  - Dermavant Investigator Site, San Antonio, Texas
  - Dermavant Investigator Site, Norfolk, Virginia
- Canada (4):
  - Surrey, British Columbia
  - Dermavant Investigator Site, Richmond, Ontario
  - Dermavant Investigator Site, Waterloo, Ontario
  - Dermavant Investigational Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided